CLINICAL TRIAL: NCT04217577
Title: Dried Plum Supplementation as Treatment for Bone Loss Following Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Restriction on in-person research due to COVID-19
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Beatrice Jenny Kiratli PhD, Research Health Scientist, VA Palo Alto Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KIB0033
Record Dates: First submitted 2019-12-30; First posted 2020-01-03 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dried Plums (Experimental): Consume dried plums daily.
  Interventions: Dietary Supplement: Dried plums

INTERVENTIONS:
Dietary Supplement: Dried plums — 10-16 dried plums/day, approximately 100-120 g/day

SUMMARY:
The purpose of this pilot study is to explore whether dried plum (prunes) added to the diet is effective in reducing or reversing bone loss following spinal cord injury (SCI). The investigators will look for changes in bone mineral density as well as evidence in the blood of markers of bone activity. The first part of the study is to check whether participants with SCI can and will eat the required amount of dried plums (prunes) on a daily basis. The second part of the study is to follow participants over one year and look for changes in bone mass and blood markers.

DETAILED DESCRIPTION:
Recruitment & screening: SCI clinicians will invite patients from the VA SCI Center census to participate in the pilot in person during a clinic visit or inpatient admission. If the patient is interested, one of the study team will explain the study and obtain consent. The study will be performed on an outpatient basis with return to the VA for study visits at 3, 6 ,9 , and 12 months.

The investigators will mail Opt-Out Letters to individuals who have been identified as potentially eligible. The Opt-Out Letter will include a Response Letter and a Return Self-addressed Stamped Envelope (attached). If the investigators do not receive a NO response by phone or mail after 2 weeks, they will attempt to call using an Opt-Out Telephone Script and Recruitment Script (Attached).

Screening is primarily done based on interest, medical history and contraindications. There may be blood values, collected at baseline that indicate ineligibility, but these will be determined on individual cases. Interest in the study and commitment to maintain the study diet/intake will be important to ascertain - although the investigators anticipate that there may be dropout or reduced compliance with time.

Procedures:

1. For the first month, each participant will consume 6-8 prunes per day to determine tolerability. Starting in Month 2, each participant will consume approximately 10-16 prunes/day (<120 g), depending on the size of the prune. The smaller prunes weigh about 7 g and the larger weigh up to 10 g. It will be suggested to consume 5-8 prunes twice per day for breakfast and dinner. However, this is not a requirement, so long as the per-day goal is met. If a participant does not eat the daily requirement one day they will be encouraged to make up the difference over the next 6 days such that the total is equal to the required 100-112 total prunes for the week. If however, they miss multiple days of prune consumption, they will be asked to contact the study coordinators to develop a reasonable plan to get back on track.
2. Participants will be asked to track consumption regularly by use of a chart. They will be instructed to note days when they missed or consumed fewer prunes. They will also be instructed to note any changes in bowel or other function and contact study staff with any questions.

Assessments:

1. Bone mineral density by dual xray absorptiometry (DXA) to include the following sites: total body, spine, bilateral hip, bilateral knee. Total body scans will be obtained at baseline and at 12 months; all other scans will be obtained at baseline, 3, 6, 9, and 12 months.
2. Blood assessments will be collected at the same intervals and will include serum concentrations of C-terminal telopeptide (CTX), which is a bone resorption marker, and Procollagen Type I Intact N-Terminal Propeptide (P1NP), a bone formation marker to measure the rate and direction of bone metabolism during the study. Serum will be frozen for batch processing. Safety labs will also be drawn including a comprehensive metabolic panel, primarily to monitor renal function, calcium concentration, and blood sugar. Magnesium and phosphorus levels will also be analyzed. De-identified, coded blood samples will be sent to Quest Diagnostics Lab (contracting lab) for analysis.
3. Surveys will be administered to the participants at 0, 3, 6, 9, and 12 months. These will include the Global Health Scale- to evaluate overall health and well-being, the Spinal Cord Injury Quality of Life Questionnaire (SCI-QOL) on Bowel Management as well as the Bristol Stool Chart-to ascertain any affects the consumption of prunes have on participants' bowel habits. Finally participants will be given a brief questionnaire regarding their activity level, general health status, lifestyle habits, and participation characteristics while in the study.

Study Contact: For the first month, study staff will call each participant weekly to ask about any concerns or issues related to prune consumption. After this, calls will be less frequent, biweekly for the next month(s) and once per month after this. As this is a pilot study, the investigators may adjust the call frequency as needed to determine if more or fewer calls are needed. One of the main goals of this pilot is to determine feasibility related to regular consumption; the investigators feel that useful information can be gathered by calling rather than waiting for the participant to contact us.

ELIGIBILITY:
Inclusion Criteria:

* SCI at any level, America Spinal injury Association (ASIA) Impairment Scale = A-C
* Primarily wheelchair-user
* Age - between 18 and 65 years old.
* Two cohorts will be recruited:

  1. chronic injury greater than 4 yr and
  2. newly injured, less than 4 years
* The investigators will target Vit D blood level to be 20 ng/ml or higher and suggest that any potential participants with Vit D greater than 10 but below 20 receive a clinical protocol to achieve 20 ng/ml.

Exclusion Criteria:

* Presence of hyper/hypo-parathyroidism, renal insufficiency (GFR<60ml/min), currently taking hormone replacement therapy, severe vitamin D deficiency (<10 ng/ml), thyroid disease, active cancer diagnosis, currently using bisphosphonate or parathyroid hormone therapy, diagnosed fracture less than 3 months ago, current pressure sore stage III or IV, New York Heart Association (NYHA) functional classification of stage II-IV, inflammatory bowel disease, cirrhosis of the liver, consuming more than 3 dried plums/day as their regular diet.
* Vitamin D blood level below 10 ng/ml

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Change in Procollagen Type I Intact N-Terminal Propeptide (P1NP) | change from baseline to 12 months
  Blood marker of bone formation
Change in C-terminal telopeptide (CTX) | change from baseline to 12 months
  Blood marker of bone resorption
Change in Bone mineral density (BMD) - multiple sites | change from baseline to 12 months
  BMD of hip and knee

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is very preliminary and we are not sure yet if sharing will be valuable as we may make protocol amendments depending on study data.